CLINICAL TRIAL: NCT01630759
Title: Remote Monitoring of Diabetes in Pregnancy: a Feasibility Study for a Randomised Controlled Trial
Brief Title: Remote Monitoring of Diabetes in Pregnancy: a Feasibility Study
Acronym: Tele-Mum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Western Health and Social Care Trust (Other); Letterkenny General Hospital (Other Government); University College Hospital Galway (Other)
Responsible Party: Principal Investigator, Professor Vivien Coates, Professor, University of Ulster
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11/0016; 11/NI/0023 (Other: ORECNI)
Record Dates: First submitted 2012-06-22; First posted 2012-06-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Gestational Diabetes
Keywords: Gestational diabetes; telemonitoring; telehealth; feasibility study
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemonitoring (Experimental): The telemonitoring group will receive usual care but be asked to download their blood sugar readings and take a blood pressure and weight measurement each week. This will be reviewed by their diabetes health care team to assess the possibility of replacing alternate anti-natal/diabetes clinics with telemonitoring review in a future study. Acceptability to staff and patients will be assessed through a questionnaire (patients only) and qualitative interviews.
  Interventions: Device: Telemonitoring
- Control group (Active Comparator): Control group will consist of usual care and review at clinic.
  Interventions: Other: Control

INTERVENTIONS:
Device: Telemonitoring — Use of telemonitoring facilities to monitor weight, blood pressure and blood sugar during pregnancy complicated by gestational diabetes
  Arms: Telemonitoring
Other: Control — The control group will receive usual diabetes/antinatal care. The outcomes from usual care will be compared with the outcomes from the telemonitoring group in order to ensure that it provides comparable care.
  Other Names: Usual care
  Arms: Control group

SUMMARY:
When women with diabetes become pregnant it is particularly important to control blood sugar levels to prevent complications. Women are advised to test their blood glucose levels seven times a day and to attend antenatal and diabetes clinics every 1-2 weeks throughout the pregnancy. For those living in rural areas in the North and West of Ireland getting to a hospital specialising in the management of diabetes and pregnancy on such a regular basis can be a challenge.

Telemonitoring provides a possible solution to this problem by allowing patients to monitor their vital signs at home and transmit the information via telephone to their healthcare provider. If women could be safely monitored remotely for every other appointment it would mean that they would only need to visit the hospital once a month on a routine basis but with the option of attending the hospital if the remote telemonitoring indicated that this were necessary.

The aim of this study is to assess the feasibility and the acceptability of using remote telemonitoring facilities between antenatal women with gestational diabetes and the diabetes team and the possibility of replacing alternate diabetic review clinics with remote telemonitoring. In addition this study will explore the feasibility of running a full randomised control trial of this topic.

Women will be asked to monitor their blood sugar levels seven times a day which is part of usual care. However those in the remote telemonitoring group will be asked to measure their blood sugar using a meter that can transmit the results via a telephone line and to transmit them weekly. They will also be asked to measure their blood pressure and weight weekly and to download these results weekly for a health care professional to review. These results will be reviewed on a weekly basis by a health care professional who will contact the patient if necessary to discuss the results. Women will be followed-up from the date of diagnosis through to delivery.

Both staff and patients will be asked to give their views on the safety and acceptability of remote telemonitoring through questionnaires, focus groups or interviews. The management decisions made on reviewing the intervention group in clinic and reviewing remote telemonitoring results will also be recorded. In order for remote telemonitoring to be a viable replacement for clinic review it must allow health care professionals to make comparable management decisions. Clinical data will be collected in order to provide descriptive statistics for those who take part and to ensure that this information could be collected in any future Randomised Control Trial (RCT) looking at this topic.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Gestational Diabetes or IGT following an oral glucose tolerance test performed at the 24-28 week screening appointment
* Able to use the telehealth equipment following training by staff from the company providing telehealth services
* Have sufficient communication skills [hearing, speech & language] to be fully involved.
* Willing to use one of the approved blood glucose meters for self monitoring of blood glucose, for the duration of the study.

Exclusion Criteria:

* Previously diagnosed Type 1 diabetes or Type 2 diabetes as evidenced by medical records.
* Other diagnosed medical problems or medical therapy such as steroid therapy that would influence blood glucose control and to be decided by the endocrinologist prior to recruitment. Such exclusions to be noted by the endocrinologist or diabetes nurse specialist.
* Previous gestational diabetes is not an exclusion criterion.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | At 36-39 weeks gestation
  The previously validated 'Telemedicine satisfaction and usefulness questionnaire' will be used to assess patient satisfaction with the telemonitoring service.
  Qualitative interviews exploring the patient experience of telemonitoring will also be carried out and then analysed using the framework approach. An adapted version of this questionnaire looking specifically at the use of a blood glucose meter will be given to the control group.
Health care staff satisfaction | At completion of the study estimated to be January 2013
  The professionals involved in caring for the women using remote telemonitoring technology in antenatal or diabetes clinics will be invited to take part in a focus group at each site. If it is not possible to arrange a time and place suitable for staff in order to hold a focus group it may be necessary to hold one to one structured interviews with staff. The questions used in the focus group will aim to assess the acceptability of telemonitoring to health care staff who use it.
Management decision comparison | At weekly clinic or telemonitoring review from time recruited into study to delivery, estimated at an average of twelve weeks.
  Weighted kappa will be used to meaure the level of agreement in between clinic and telemonitoring review management decisions (in excess of the amount of agreement that we would expected by chance). This will allow the determination of inter-rater, intra-rater and inter-institutional agreement between clinic and telemonitoring review management decisions.

SECONDARY OUTCOMES:
HbA1c | Monthly for duration of participation in study, estimated at 2-3 months
  HbA1c mmol/l and IFCC units
Mean fasting blood glucose | Weekly for duration of participation in study, estimated at 12 weeks
  mmol/l plasma glucose
Blood pressure | Weekly for duration of participation in study, estimated at 12 weeks
  mmHg
Gestational age at delivery | At delivery
  Gestational age in weeks at delivery
Type of delivery | At delivery
  Vaginal or Caesarean section
Pre-eclampsia | At delivery
  Presence or absence of any pre-eclampsia
Documented problems with pregnancy | At delivery
  Presence of any documented problems during pregnancy
Weight of baby | At birth
  Weight in kg
Apgar score | At birth
  Apgar score at one and five minutes (out of 10)
Admission to neonatal unit | At one day after birth
  Whether the baby needed admission to the neonatal unit
Respiratory distress | At one day after birth
  Presence of any episodes of documented Respiratory distress in first 24 hours of life
Jaundice | At one day after birth
  Presence of any jaundice in first 24 hours of life
Neonatal hypoglycaemia | At one day after birth
  Presence of any documented episodes of neonatal hypoglycaemia in first 24 hours of life
Shoulder dystocia | At birth
  Presence of any shoulder dystocia
Malformations | At delivery
  Any malformations at delivery
Post-prandial blood glucose | Weekly for duration of participation in study, estimated at 12 weeks
  mmol/l plasma glcuose
Length of baby | At birth
  centimeters
Macrosomia | At birth
  Presence or absence of macrosomia
Head circumference | At birth
  centimeters
Average number of monitoring episodes per day | At delivery
  Average number of monitoring episodes per day
Number of downloads missed | At delivery
  Number of downloads missed by those in the telemonitoring group

CONTACTS AND LOCATIONS:
Overall Officials: Vivien E Coates, PhD, Principal Investigator — University of Ulster
Locations (2):
- Letterkenny General Hospital, Letterkenny, Donegal, Ireland
- Altnagelvin Hospital, Londonderry, Londonderry, United Kingdom

REFERENCES:
- [Derived] Given JE, Bunting BP, O'Kane MJ, Dunne F, Coates VE. Tele-Mum: A Feasibility Study for a Randomized Controlled Trial Exploring the Potential for Telemedicine in the Diabetes Care of Those with Gestational Diabetes. Diabetes Technol Ther. 2015 Dec;17(12):880-8. doi: 10.1089/dia.2015.0147. Epub 2015 Sep 22. PMID 26394017